CLINICAL TRIAL: NCT00384904
Title: Open-Label, Multiple-Dose, Drug Interaction Study to Assess the Effect of Famotidine With or Without Tenofovir on the Pharmacokinetics of Atazanavir When Given With Ritonavir in HIV-Infected Subjects
Brief Title: Drug Interaction Study of Famotidine and Atazanavir With Ritonavir in HIV-Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-328
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2008-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — atazanavir, ritonavir drug combination; Atazanavir Sulfate; Ritonavir; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A1 (No Intervention)
  Interventions: Drug: Atazanavir/Ritonavir
- A2 (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir + Famotidine
- A3 (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir + Famotidine
- B1 (No Intervention)
  Interventions: Drug: Atazanavir/Ritonavir
- B2 (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir + Tenofovir Disproxil Fumrarate + Famotidine
- B3 (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir + Tenofovir Disproxil Fumrarate + Famotidine

INTERVENTIONS:
Drug: Atazanavir/Ritonavir — Capsules/capsules, Oral, 300/100 mg, Once daily, 10 days.
  Other Names: Reyataz
  Arms: A1
Drug: Atazanavir/Ritonavir + Famotidine — Capsules/capsules + Tablets, Oral, 300/100 mg + 40 mg, Once daily + Twice daily, 7 days.
  Other Names: Reyataz
  Arms: A2
Drug: Atazanavir/Ritonavir + Famotidine — Capsules/capsules + Tablets, Oral, 300/100 mg + 20 mg, Once daily + Twice daily, 7 days.
  Other Names: Reyataz
  Arms: A3
Drug: Atazanavir/Ritonavir — Capsules/capsules + Tablets, Oral, 300/100 mg, Once daily, 10 days.
  Other Names: Reyataz
  Arms: B1
Drug: Atazanavir/Ritonavir + Tenofovir Disproxil Fumrarate + Famotidine — Capsules/capsules + Tablets + Tablets, Oral, 300/100 mg + 300 mg + 40 mg, Once daily + Twice daily, 7 days.
  Other Names: Reyataz
  Arms: B2
Drug: Atazanavir/Ritonavir + Tenofovir Disproxil Fumrarate + Famotidine — Capsules/capsules + Tablets + Tablets, Oral, 300/100 mg + 300 mg + 20 mg, Once daily + Twice daily, 7 days.
  Other Names: Reyataz
  Arms: B3

SUMMARY:
The purpose of this clinical research study is to assess the effect of Famotidine given twice daily on Atazanavir administered with Ritonavir in HIV-Infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected male and female subjects between the ages of 18 to 65 years old with a BMI 18 to 35 kg/m²
* Prior to enrollment subjects must be currently receiving Atazanavir/Ritonavir plus at least 2 NRTIs, must have plasma HIV RNA <400 copies/mL and have CD4 count >200 cells/mm³

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Atazanavir plasma drug concentrations | on days 10, 11, 17, 18, 24 and 25

SECONDARY OUTCOMES:
Ritonavir plasma drug concentrations | on days 10, 11, 17, 18, 24 and 25
Safety measures: Physical examinations
ECGs | entry and discharge
laboratory tests including, liver and renal function | entry, discharge and days 11, 18
CD4 count | discharge
HIV viral load | entry and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (3):
  - Garden State Infectious Disease Associates, Pa, Voorhees Township, New Jersey
  - Unc Center For Aids Research, Chapel Hill, North Carolina
  - Local Institution, Philadelphia, Pennsylvania
- Local Institution, London, Greater London, United Kingdom